CLINICAL TRIAL: NCT01554332
Title: A Clinical Evaluation for the Management of Patients With Chronic Neuropathic Pain With Cortical Stimulation
Brief Title: Motor Cortex Stimulation for Chronic Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C-11-13
Record Dates: First submitted 2012-01-13; First posted 2012-03-14 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Neuropathic Pain; Facial Pain; Post-stroke Pain; Brachial Plexus Avulsion; Phantom Limb Pain of the Upper Extremities
Keywords: Motor Cortex Stimulation; Neuropathic pain
MeSH Terms: conditions — Neuralgia; Facial Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active stimulation (Active Comparator)
  Interventions: Device: Motor Cortex Stimulation using SJM EonC Stimulator
- Sham stimulation (Sham Comparator)
  Interventions: Device: Motor Cortex Stimulation using SJM EonC Stimulator

INTERVENTIONS:
Device: Motor Cortex Stimulation using SJM EonC Stimulator — Patients will be randomized to receive either active stimulation the first 3 months followed by a one-month washout, followed by Sham Stimulation the next 3 months, vs. the reverse order of treatment, followed by single blind stimulation, and an open label phase.

SUMMARY:
The purpose of this study is to evaluate the efficacy of cortical stimulation (CS) as an adjunctive treatment for chronic neuropathic pain.

DETAILED DESCRIPTION:
Prospective, controlled, double blind, randomized, crossover study with endpoint evaluations at the end of each 3-month treatment period.

An interim analysis will be conducted by a blinded committee when approximately half of the patients have finished the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (non-pregnant) age 21-70 years;
* Able to give informed consent in accordance with institutional policies;
* Diagnosis of chronic neuropathic pain according to the DN4 Neuropathic Pain Diagnosis scale (score ≥ 4).
* Documented pain for at least 12 months;
* Documented previous or current treatment for neuropathic pain with medications from at least two of the following groups at adequate doses: antidepressants, anticonvulsants, and/or gabapentinoids;
* VAS scores of at least 6 during baselines #1 and 2.
* Documented clinical diagnosis of neuropathic pain associated with one of the following conditions: facial pain, post-stroke pain, brachial plexus avulsion, or phantom limb pain of the upper extremities.
* In the group with post-stroke pain, only patients with predominant face and upper extremity pain will be included. This will be defined as a difference of ≥ 30% or ≥ 2 points in VAS scores between these regions and lower extremity (in patients who also have pain in the leg).
* No change in current neuropathic pain medication regimen for at least 4 weeks prior to study enrollment.
* Able to comply with all testing and follow-up requirements as defined by the study protocol.
* Must be determined medically stable by surgeon to undergo cortical stimulation surgical procedure.

Exclusion Criteria:

* Alcohol, medication, or illegal substance dependence or abuse within last 12 months;
* Trigeminal neuralgia or atypical facial pain.
* Post-stroke pain predominantly in the lower extremity.
* Advanced cardiovascular disease which renders anesthesia and surgery as unsafe as determined by neurosurgeon;
* Clinically relevant abnormality (e.g. tumor) on study MRI;
* Has cardiac pacemaker/defibrillator or other implanted active stimulator;
* Has a medical condition requiring a repetitive MRI body scan;
* Requires chemotherapy for the treatment of malignancy or requiring chronic oral or intravenous, immunosuppressive, or steroid therapy;
* Is unable to comply with study visit schedule and timeline;
* Past ablative or relevant intracranial surgery;
* A female lactating or of child bearing potential, with a positive pregnancy test or not using adequate contraception;
* Other medical conditions likely to require hospitalization within the next year.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-10; Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Approximately 7 months
  The primary analysis of effectiveness is based on the mean differences in changes from the period-specific baseline in VAS scores when patients are receiving 3 month of active vs. 3 months of sham stimulation on a double-blinded fashion.

SECONDARY OUTCOMES:
Visual Analog Scale, responder | Participants will be followed for approximatley 18 months
  defined as a ≥30% or 2 points reduction from baseline in VAS scores
Neuropathic Pain Symptom Inventory (NPSI) | Participants will be followed for approximatley 18 months
Brief Pain Inventory (BPI) | Participants will be followed for approximatley 18 months
Short Form of the McGill Pain Questionnaire(SF-MPQ) | Participants will be followed for approximatley 18 months
Sickness Impact Profile (SIP) | Participants will be followed for approximatley 18 months
Medication Quantification Scale (MQS) | Participants will be followed for approximatley 18 months
SF-36 Health Survey and safety | Participants will be followed for approximatley 18 months
Pain Catastrophizing Scale (PCS) | Participants will be followed for approximatley 18 months
Global Impression of Change (patient and evaluator's version) | Participants will be followed for approximatley 18 months
Device related Adverse Events | Participants will be followed for approximatley 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Karst, Study Director — Abbott Neuromodulation
Locations (1):
- University of São Paulo - Hospital das Clínicas, São Paulo, Brazil